CLINICAL TRIAL: NCT05833685
Title: Predicting Changes in Core Muscles During Female Sexual Dysfunction: A Comprehensive Analysis Using Machine and Deep Learning
Status: Completed | Type: Observational
Sponsor: Deraya University (Other)
Responsible Party: Sponsor
Other Study IDs: P.REC/ 6/2023
Record Dates: First submitted 2023-04-16; First posted 2023-04-27 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Female Sexual Dysfunction
Keywords: Core Muscles, machine learning,female sexual dysfunction, KNN

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Female sexual dysfunction group
  Interventions: Other: no intervention
- Normal females
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The purpose of this study is to Predicting changes in core muscles during female sexual dysfunction by A Comprehensive Analysis Using Machine and Deep Learning Female sexual dysfunction (FSD) is a common condition that affects womenof all ages. It is characterized by a range of symptoms, including decreased libido, difficulty achieving orgasm, and pain during intercourse. One potential cause of FSD is muscular weakness or changes in the core muscles. These muscles play an important role in sexual function, and changes in their strength or activation patterns can lead to FSD. Additionally, the development of a machine learning model for this purpose could pave the way for future studies exploring the use of artificial intelligence in the diagnosis and treatment of other musculoskeletal disorder and female health issues.

ELIGIBILITY:
Inclusion Criteria:

* a number of parities ≤ three
* normal vaginal deliveries

Exclusion Criteria:

* History of a recto-vaginal or vesico-vaginal fistula, undiagnosed uterine bleeding urinary tract infection,
* diabetes,
* intrauterine device
* sexual disorder

Ages: 30 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: 100 patients were distributed randomly into two groups. Female sexual dysfunction group and another group is normal females. Two group will be measure Transverses muscle ratio, Multifidus muscle ratio ,diaphragm excursion and force of contraction of pelvic floor muscles by ultrasound imaging, VLQ and FSFI questionnaires for female sexual function VLQ and FSFI questionnaires for female sexual dysfunction and normal females. Patients will be examined by radiologist with medical ultrasound imaging
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Diaphragm excursion | 2 months
  Ultrasound imaging curvilinear transducer

SECONDARY OUTCOMES:
Force of contraction of pelvic floor muscles | 2 months
  ultrasound imaging, convex transducer was used at a frequency of 5 MHz for evaluating. Voluntary PFM contractions' force (strength) of all patients. It has a good inter-rater reliability for measuring PFM force (ICC, 0.81, 0.7123) respectively, as well as a good intra-rater reliability (ICC,0.98, 0.9841) respectively

CONTACTS AND LOCATIONS:
Locations (1):
- Deraya university, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No